CLINICAL TRIAL: NCT02499679
Title: Assessing Diagnostic Value of Non-invasive FFRCT in Coronary CarE (ADVANCE)
Brief Title: Assessing Diagnostic Value of Non-invasive FFRCT in Coronary Care
Acronym: ADVANCE
Status: Completed | Type: Observational
Sponsor: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-905-001
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients diagnosed with CAD by cCTA: All clinically stable, symptomatic patients diagnosed with CAD by coronary computed tomography angiography (cCTA), that meet eligibility criteria, and are able and willing to participate are candidates for the ADVANCE Registry. Those patients that meet all inclusion/exclusion criteria and who sign the ethics committee (EC)/institutional review board (IRB) approved informed consent will be enrolled in the registry. FFRCT shall be used in accordance with the current Instructions for Use (IFU) document.

SUMMARY:
The objective of the HeartFlow ADVANCE Registry is to evaluate utility, clinical outcomes and resource utilization of FFRCT-guided evaluation in clinically stable, symptomatic patients with coronary artery disease (CAD) in order to further inform patients, health care providers, and other stakeholders about which technologies are most effective and efficient in the diagnosis and management of CAD.

DETAILED DESCRIPTION:
REGISTRY OBJECTIVE

The objective of the HeartFlow ADVANCE Registry is to evaluate utility, clinical outcomes and resource utilization of FFRCT-guided evaluation in clinically stable, symptomatic patients with CAD in order to further inform patients, health care providers, and other stakeholders about which technologies are most effective and efficient in the diagnosis and management of CAD.

SPECIFIC OBJECTIVES:

1. To determine if the availability of FFRCT, in addition to coronary anatomy from the cCTA, will lead to a significant change in the coronary management plan.
2. To assess the real world outcomes of utilizing FFRCT to guide invasive management and/or medical treatment.
3. To assess resource utilization, following standard practice for diagnostic and treatment pathways incorporating FFRCT as the preferred CAD diagnostic test.
4. To provide society including patients, health care providers, and other stakeholders with information about which diagnostic technologies are most effective and efficient in managing patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Clinically stable, symptomatic patients who undergo cCTA and are diagnosed with CAD and meet eligibility criteria for FFRCT.

Exclusion Criteria:

1. cCTA showing no CAD
2. Uninterpretable cCTA by site assessment, in which severe artifacts prevent angiographic evaluation
3. Any active, serious, life-threatening disease with a life expectancy of less than 1 year
4. Inability to comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All clinically stable, symptomatic patients diagnosed with CAD by cCTA, that meet eligibility criteria, and are able and willing to participate are candidates for the ADVANCE Registry. Those patients that meet all inclusion/exclusion criteria and who sign the EC/IRB approved informed consent will be enrolled in the registry. FFRCT shall be used in accordance with the current Instructions for Use document.
Sampling Method: Non-Probability Sample
Enrollment: 4737 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manesh Patel, MD, Principal Investigator — Duke Health; Jonathon Leipsic, MD, Principal Investigator — Providence Health & Services; Koen Nieman, MD, Principal Investigator — Erasmus Medical Center; Takashi Akasaka, MD, Principal Investigator — Wakayama Medical University

REFERENCES:
- [Derived] Dundas J, Leipsic J, Fairbairn T, Ng N, Sussman V, Guez I, Rosenblatt R, Hurwitz Koweek LM, Douglas PS, Rabbat M, Pontone G, Chinnaiyan K, de Bruyne B, Bax JJ, Amano T, Nieman K, Rogers C, Kitabata H, Sand NPR, Kawasaki T, Mullen S, Huey W, Matsuo H, Patel MR, Norgaard BL, Ahmadi A, Tzimas G. Interaction of AI-Enabled Quantitative Coronary Plaque Volumes on Coronary CT Angiography, FFRCT, and Clinical Outcomes: A Retrospective Analysis of the ADVANCE Registry. Circ Cardiovasc Imaging. 2024 Mar;17(3):e016143. doi: 10.1161/CIRCIMAGING.123.016143. Epub 2024 Mar 12. PMID 38469689
- [Derived] Gulsin GS, Tzimas G, Holmes KR, Takagi H, Sellers SL, Blanke P, Koweek LMH, Norgaard BL, Jensen J, Rabbat MG, Pontone G, Fairbairn TA, Chinnaiyan KM, Douglas PS, Huey W, Matsuo H, Sand NPR, Nieman K, Bax JJ, Amano T, Kawasaki T, Akasaka T, Rogers C, Berman DS, Patel MR, De Bruyne B, Mullen S, Leipsic JA. Impact of Coronary CT Angiography-derived Fractional Flow Reserve on Downstream Management and Clinical Outcomes in Individuals with and without Diabetes. Radiol Cardiothorac Imaging. 2023 Oct 19;5(5):e220276. doi: 10.1148/ryct.220276. eCollection 2023 Oct. PMID 37908552
- [Derived] Madsen KT, Norgaard BL, Ovrehus KA, Jensen JM, Parner E, Grove EL, Fairbairn TA, Nieman K, Patel MR, Rogers C, Mullen S, Mickley H, Rohold A, Botker HE, Leipsic J, Sand NPR. Prognostic Value of Coronary CT Angiography-derived Fractional Flow Reserve on 3-year Outcomes in Patients with Stable Angina. Radiology. 2023 Sep;308(3):e230524. doi: 10.1148/radiol.230524. PMID 37698477
- [Derived] Fairbairn TA, Dobson R, Hurwitz-Koweek L, Matsuo H, Norgaard BL, Ronnow Sand NP, Nieman K, Bax JJ, Pontone G, Raff G, Chinnaiyan KM, Rabbat M, Amano T, Kawasaki T, Akasaka T, Kitabata H, Binukrishnan S, Rogers C, Berman D, Patel MR, Douglas PS, Leipsic J. Sex Differences in Coronary Computed Tomography Angiography-Derived Fractional Flow Reserve: Lessons From ADVANCE. JACC Cardiovasc Imaging. 2020 Dec;13(12):2576-2587. doi: 10.1016/j.jcmg.2020.07.008. Epub 2020 Aug 26. PMID 32861656
- [Derived] Pontone G, Weir-McCall JR, Baggiano A, Del Torto A, Fusini L, Guglielmo M, Muscogiuri G, Guaricci AI, Andreini D, Patel M, Nieman K, Akasaka T, Rogers C, Norgaard BL, Bax J, Raff GL, Chinnaiyan K, Berman D, Fairbairn T, Koweek LH, Leipsic J. Determinants of Rejection Rate for Coronary CT Angiography Fractional Flow Reserve Analysis. Radiology. 2019 Sep;292(3):597-605. doi: 10.1148/radiol.2019182673. Epub 2019 Jul 23. PMID 31335283
- [Derived] Patel MR, Norgaard BL, Fairbairn TA, Nieman K, Akasaka T, Berman DS, Raff GL, Hurwitz Koweek LM, Pontone G, Kawasaki T, Sand NPR, Jensen JM, Amano T, Poon M, Ovrehus KA, Sonck J, Rabbat MG, Mullen S, De Bruyne B, Rogers C, Matsuo H, Bax JJ, Leipsic J. 1-Year Impact on Medical Practice and Clinical Outcomes of FFRCT: The ADVANCE Registry. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 1):97-105. doi: 10.1016/j.jcmg.2019.03.003. Epub 2019 Mar 17. PMID 31005540
- See also: Real-world clinical utility and impact on clinical decision-making of coronary computed tomography angiography-derived fractional flow reserve: lessons from the ADVANCE Registry — https://pubmed.ncbi.nlm.nih.gov/30165613/
- See also: 1-Year Impact on Medical Practice and Clinical Outcomes of FFRCT: The ADVANCE Registry — https://doi.org/10.1016/j.jcmg.2019.03.003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All clinically stable, symptomatic patients diagnosed with CAD by coronary CTA that meet the following eligibility criteria are candidates for enrollment in the ADVANCE Registry: age >18 years, ability to provide informed consent, and meet eligibility criteria for FFRCT based on CAD, with an anatomical stenosis >25%, diagnosed on coronary CTA.
Pre-assignment Details: The ADVANCE Registry screened a total of 5,083 patients, and 4,893 of them had coronary CTA submitted for FFRCT analysis. Of these submitted, 4,737 (96.80%) were of sufficient image quality for FFRCT analysis.
Groups:
- All Patients Diagnosed With CAD by cCTA+FFRCT: All clinically stable, symptomatic patients diagnosed with CAD by coronary computed tomography angiography (cCTA) and FFRCT (Fractional Flow Reserve derived from coronary computed tomography angiography).
Period: Overall Study
Arm/Group | All Patients Diagnosed With CAD by cCTA+FFRCT
Started | 4737
Completed | 4737
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There was no significant difference between subject group demographics or risk factors for those receiving CCTA alone vs. CCTA plus FFRCT. Information represented in this table is for all subjects with FFRCT results and data available.
Groups:
- Patients Diagnosed With CAD by cCTA: All clinically stable, symptomatic patients diagnosed with CAD by coronary computed tomography angiography (cCTA), that meet eligibility criteria, and are able and willing to participate are candidates for the ADVANCE Registry. Those patients that meet all inclusion/exclusion criteria and who sign the ethics committee (EC)/institutional review board (IRB) approved informed consent will be enrolled in the registry.
  Obstructive CAD will be defined as luminal diameter stenosis >50% by invasive angiography visual assessment or non-invasive cCTA, or invasively measured FFR of ≤0.80.
  cCTA is defined as coronary computed tomographic angiography. FFR (Fractional Flow Reserve) is defined as the ratio of the mean distal intracoronary arterial pressure, (Pd) to the mean arterial pressure (Pa) under conditions of adenosine induced maximal hyperemia.
Arm/Group | Patients Diagnosed With CAD by cCTA
Number analyzed (Participants) | 4737
Age, Continuous [Mean (Standard Deviation); unit: years] — There was no significant difference between subject group demographics or risk factors for those receiving CCTA alone vs. CCTA plus FFRCT. Information represented in this table is for all subjects with FFRCT results. Population: There was no significant difference between subject group demographics or risk factors for those receiving CCTA alone vs. CCTA plus FFRCT. Information represented in this table is for all subjects with FFRCT results.
  years | 66.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There was no significant difference between subject group demographics or risk factors for those receiving CCTA alone vs. CCTA plus FFRCT. Information represented in this table is for all subjects with FFRCT results.
  Participants
    Female | 1603
    Male | 3134
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 3045
Diabetus mellitus [Count of Participants; unit: Participants] | 1136
Hyperlipidemia [Count of Participants; unit: Participants] | 2957
Smoking [Count of Participants; unit: Participants]
  Current smoking | 797
  Former smoker | 1615
  Never smoked | 1973
  Unknown | 352
Angina status [Count of Participants; unit: Participants] — Population: There was no significant difference between subject group demographics or risk factors for those receiving CCTA alone vs. CCTA plus FFRCT. Information represented in this table is for all subjects with FFRCT results.
  Participants
    Atypical | 1727
    Typical | 1025
    Non-cardiac pain | 297
    Dyspnea | 472
    None | 1164
    Unknown | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reclassification of CAD Management, Assessed as the Therapeutic Recommendations Made Based on Review of Coronary CTA Alone Versus CTA + FFRCT, When Available, by a Central Integration Core Laboratory.
Description: The reclassification rate of management plans was assessed by the blinded independent review committee and local physician teams separately. These evaluations are meant to assess the potential impact of FFRCT on downstream testing and clinical decision making but were not be used to determine actual patient care. This endpoint is aimed at determining the incremental value of FFRCT over coronary CTA alone in the management of stable angina.
  FFRCT is non-invasive method to determine FFR which computes the hemodynamic significance of CAD (FFRCT) from subject-specific cCTA data using computational fluid dynamics under rest and simulated maximal coronary hyperemic conditions (Taylor 2013).
Time Frame: at 90 days
Population: The primary endpoint of reclassification between core lab CCTA alone and CCTA plus FFRCT-based management.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Reclassification Rate by Core Lab: For each enrolled patient, the endpoint review committee used data from coronary CTA and FFRCT, along with the clinical data such as medical history and demographics to determine the management plan using the following criteria: (a) optimal medical therapy, (b) percutaneous coronary intervention, (c) coronary artery bypass graft surgery, or (d) more information required. The management plan recommended by the committee was compared with the therapy that the patient received, as determined by his or her local team of physicians.
Arm/Group | Reclassification Rate by Core Lab
Number analyzed (Participants) | 4737
percentage of participants | 66.9 [64.8 to 67.6]

2. Secondary Outcome: Percentage of Participants With Reclassification Between Investigator Management Plan Based on cCTA Alone Compared to Actual Clinical Management
Description: Coronary computed tomography angiography-derived fractional flow reserve resulted in revision of the clinical management plan as determined by the site investigators.
Time Frame: at 90 days
Population: All participants who were enrolled in the study and received cCTA and FFRCT analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Reclassification Rate by Investigator Management Plan: For each enrolled patient, investigators used data from coronary CTA and FFRCT, along with the clinical data such as medical history and demographics to determine the management plan using the following criteria: (a) optimal medical therapy, (b) percutaneous coronary intervention, (c) coronary artery bypass graft surgery, or (d) more information required. The management plan recommended by investigator was compared with the therapy that the patient received, as determined by his or her local team of physicians.
Arm/Group | Reclassification Rate by Investigator Management Plan
Number analyzed (Participants) | 4737
percentage of participants | 63.5 [62.0 to 65]

3. Secondary Outcome: Percentage of Participants With Invasive Catheterization Without Obstructive Disease
Description: Invasive catheterization without obstructive disease was measured by either site read coronary angiogram showing no stenosis of ≥ 50% or no invasively-measured FFR ≤ 0.80 in a segment distal to a stenosis.
Time Frame: At 90 days
Population: The rate of anatomically defined 'non-obstructive' disease at ICA (no stenosis defined as >50% at ICA)
Measure: Number; unit: percentage of participants
Groups:
- ICA Patients With FFRCT >0.80: Patients undergoing ICA procedure and FFRCT result showing Non-Obstructive CAD.
- ICA Patients With FFRCT ≤0.80: Patients undergoing ICA procedure and FFRCT result showing Obstructive CAD.
Arm/Group | ICA Patients With FFRCT >0.80 | ICA Patients With FFRCT ≤0.80
Number analyzed (Participants) | 281 | 694
percentage of participants | 43.8 | 14.4

4. Secondary Outcome: Percentage of Major Adverse Coronary Events (MACE) at 90 Days
Description: MACE is defined as the composite rate of all cause death, non-fatal myocardial infarction (MI) and unplanned hospitalization for acute coronary syndrome (ACS) leading to urgent revascularization.
Time Frame: 90 days
Population: MACE: Major adverse cardiac event (MI, Death, Hospitalization for ASC and urgent revascularization).
Measure: Count of Participants; unit: Participants
Groups:
- MACE Events Within 90 Days Subject Whose FFRCT Was >0.80: All patients who received cCTA and FFRCT. Subject whose FFRCT was >0.80 (n= 1592).
- MACE Events Within 90 Days. Patients With at Least One FFRCT Value ≤ 0.80: All patients who received cCTA and FFRCT. Subjects with at least one FFRCT value ≤ 0.80
Arm/Group | MACE Events Within 90 Days Subject Whose FFRCT Was >0.80 | MACE Events Within 90 Days. Patients With at Least One FFRCT Value ≤ 0.80
Number analyzed (Participants) | 1592 | 3145
Participants | 0 | 19

5. Secondary Outcome: Percentage of Individual Components of MACE at 90 Days
Description: Individual components of MACE defined as all cause death, non-fatal MI, unplanned hospitalization for ACS leading to urgent revascularization
Time Frame: 90 days
Population: MI - myocardial infarction ACS - acute coronary syndrome
Measure: Count of Participants; unit: Participants
Groups:
- Patients With cCTA and FFRCT > 0.80: All patients who received cCTA and FFRCT and whose FFRCT > 0.80.
- Patients With cCTA and at Least One FFRCT Value ≤ 0.80: All patients who received cCTA and FFRCT and with at least one FFRCT value ≤ 0.80
Arm/Group | Patients With cCTA and FFRCT > 0.80 | Patients With cCTA and at Least One FFRCT Value ≤ 0.80
Number analyzed (Participants) | 1592 | 3145
Participants
  MI | 0 | 4
  Urgent unplanned hospitazation for ACS and urgent revascularization. | 0 | 5
  Death | 0 | 10

6. Secondary Outcome: Cumulative Radiation Exposure From cCTA MilliSievert (mSv)
Description: Cumulative radiation exposure calculated in non-invasive coronary diagnostic tests: cCTA effective radiation dose. Effective radiation dose measured as the product of dose-length product times for conversion coefficient for the chest (K = 0.026 mSv/mGy·cm).
Time Frame: Baseline
Population: All patients referred for clinical consecutive coronary CT angiography who had FFRCT analysis performed
Measure: Mean (Standard Deviation); unit: mSv
Groups:
- All Patients Diagnosed With CAD by cCTA Undergoing cCTA and FFRCT Analysis: CAD - coronary artery disease. cCTA - coronary computed tomography angiography. FFRCT - FFR derived from coronary CT angiography,
Arm/Group | All Patients Diagnosed With CAD by cCTA Undergoing cCTA and FFRCT Analysis
Number analyzed (Participants) | 2778
mSv | 10.0 (9.1)

7. Secondary Outcome: Resource Utilization at 90 Days. Site-determined Post FFRCT Treatment Plan
Description: Resource utilization composite defined as the composite of invasive diagnostic and therapeutic coronary procedures and noninvasive cardiac testing. Site treating physician recommended clinical management strategies following coronary computed tomography angiography-derived fractional flow reserve.
Time Frame: 90 days
Population: All stable patients who undergo cCTA and are diagnosed with CAD.
Measure: Count of Participants; unit: Participants
Groups:
- Site-determined Post-FFRCT Treatment Plan - Revascularization; Site-determined Post-FFRCT Treatment Plan - Medications; Site-determined Post-FFRCT Treatment Plan - Further Diagnostics: All clinically stable, symptomatic patients diagnosed with CAD by coronary computed tomography angiography (cCTA) and FFRCT.
Arm/Group | Site-determined Post-FFRCT Treatment Plan - Revascularization | Site-determined Post-FFRCT Treatment Plan - Medications | Site-determined Post-FFRCT Treatment Plan - Further Diagnostics
Number analyzed (Participants) | 1418 | 2679 | 121
Participants
  Medical Therapy | 504 | 2545 | 92
  PCI | 799 | 115 | 25
  CABG | 115 | 19 | 4

8. Secondary Outcome: Percentage of Major Adverse Coronary Events (MACE) at 1 Year
Description: as for outcome 4
Time Frame: 1 year
Population: MACE: Major adverse cardiac event (MI, Death, Hospitalization for ASC and urgent revascularization).
Measure: Count of Participants; unit: Participants
Groups:
- MACE Events at 1 Year Subject Whose FFRCT Was >0.80: All patients who received cCTA and FFRCT. Subject whose FFRCT was >0.80 (n= 1592).
- MACE Events at 1 Year. Patients With at Least One FFRCT Value ≤ 0.80: All patients who received cCTA and FFRCT. Subjects with at least one FFRCT value ≤ 0.80
Arm/Group | MACE Events at 1 Year Subject Whose FFRCT Was >0.80 | MACE Events at 1 Year. Patients With at Least One FFRCT Value ≤ 0.80
Number analyzed (Participants) | 1592 | 3145
Participants | 12 | 43

9. Secondary Outcome: Percentage of Individual Components of MACE at 1 Year
Description: as for outcome 5
Time Frame: 1 year
Population: MI - myocardial infarction ACS - acute coronary syndrome
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With cCTA and FFRCT > 0.80 | Patients With cCTA and at Least One FFRCT Value ≤ 0.80
Number analyzed (Participants) | 12 | 43
Participants
  Death | 7 | 28
  MI | 3 | 9
  ACS leading to unplanned hospitalization and revascularization | 2 | 6

ADVERSE EVENTS:
Time Frame: Clinical Events at 1 year
Description: Note: this study involved prospective data collection to validate in a blinded manner a non-invasive test and further patient management therefore adverse event information is reported based only on the standard of care index procedure.
Groups:
- Patients Receiving cCTA and FFRCT >0.80; Patients Receiving cCTA and FFRCT≤0.80: All clinically stable, symptomatic patients diagnosed with CAD by coronary computed tomography angiography (cCTA) and received FFRCT analysis results.
Arm/Group | Patients Receiving cCTA and FFRCT >0.80 | Patients Receiving cCTA and FFRCT≤0.80
All-Cause Mortality (participants affected / at risk) | 7/4737 | 28/4737
Serious Adverse Events (participants affected / at risk) | 12/4737 | 43/4737
Other Adverse Events (participants affected / at risk) | 80/1591 | 1036/3137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving cCTA and FFRCT >0.80 (N=4737) | Patients Receiving cCTA and FFRCT≤0.80 (N=4737)
Death (any cause) (Cardiac disorders) | 7 (35) | 28 (35)
MI (Cardiac disorders) | 3 (12) | 9 (12) — MI - myocardial infarction
ACS leading to urgent hospitalization and revascularization (Cardiac disorders) | 2 (8) | 6 (8) — ACS - acute coronary syndrome
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving cCTA and FFRCT >0.80 (N=1591) | Patients Receiving cCTA and FFRCT≤0.80 (N=3137)
Revascularization (Cardiac disorders) | 80 (80) | 1036 (1036) — Revascularization: CABG - coronary artery bypass graft, PCI - percutaneous coronary intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT02499679/Prot_SAP_000.pdf